CLINICAL TRIAL: NCT02767050
Title: Incidence of Caries in Smoking and Smokeless Tobacco-An Observation Study
Brief Title: Incidence of Caries in Smoking and Smokeless Tobacco
Acronym: ICSSLT
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.Alekhya, Resident, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: PMVIDS&RC/IEC/OMR/PR/0046-15
Record Dates: First submitted 2016-02-15; First posted 2016-05-10 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: DENTAL CARIES
Keywords: DENTAL CARIES; TOBACCO USERS; SMOKERS; SMOKELESS TOBACCO CHEWERS
MeSH Terms: conditions — Dental Caries; Tobacco Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GROUP 1: CONTROL GROUPS: Patients with no habit history of tobacco are included in group 1.
- GROUP 2: SMOKING TOBACCO: Patients with a history of tobacco consumption in the form of smoking.
- GROUP 3: SMOKELESS TOBACCO: Patients with a history of tobacco consumption in the form of chewing.

SUMMARY:
The following observational study evaluates incidence of caries in smoking and smokeless tobacco based on habit history by clinical examination and DMFT index.

DETAILED DESCRIPTION:
Dental caries is an irreversible microbial disease of the calcified tissues of the teeth, characterized by demineralization of the inorganic portion and destruction of the organic substance of the tooth, which often leads to cavitation. It is a complex and dynamic process where a multitude of factors influence and initiate the progression of disease. There are practically no geographic areas in the world whose inhabitants do not exhibit some evidence of dental caries. It affects persons of both genders in all races, all socioeconomic strata and every age group. Likewise, there is strong evidence that tobacco use has numerous negative effects on oral health, for example staining of teeth, dental restoration, development of oral diseases. A biologically reasonable explanation for an association between chewing tobacco use and dental caries may be the presence of higher levels of fermentable sugars in chewing tobacco products which can stimulate the growth of carcinogenic bacteria. The decreased buffering effect possible lower pH of smokers saliva and higher number of lactobacilli and streptococcus mutans group may indicate an increased susceptibility to caries in smokers. On the other hand, there are researches which conclude that presence of extrinsic tobacco stains appear to provide a protective effect from caries.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients who are willing for the study.
* A positive history of dental caries in smokers and smokeless tobacco.
* Patients with caries not under any treatment of the same.

EXCLUSION CRITERIA:

* Unwilling patients who do not want to be a part of the study.
* Patient with fluorosis.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending Panineeya Institute of Dental Sciences and Research Centre having tobacco chewing and smoking habits without fluorosis would be included in the study after their informed consent.
  DMFT index is scored for 613 patient of both the genders, visiting OPD of oral medicine and radiology after the clinical diagnosis of caries along with radiographs. The clinical scores are recorded along with investigations and a proforma would include the habit with duration, frequency, area of placement and form of tobacco intake.
Sampling Method: Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Dental caries in smoking and smokeless tobacco chewers is determined by proper clinical examination of caries and is scored by DMFT index in both smoking and smokeless tobacco chewers separately and measured. | 5-6 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: NALLAN CHAITANYA, MDS, Principal Investigator — Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre
Locations (1):
- Panineeya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vellappally S, Jacob V, Smejkalova J, Shriharsha P, Kumar V, Fiala Z. Tobacco habits and oral health status in selected Indian population. Cent Eur J Public Health. 2008 Jun;16(2):77-84. doi: 10.21101/cejph.a3448. PMID 18661810
- [Result] Vellappally S, Fiala Z, Smejkalova J, Jacob V, Shriharsha P. Influence of tobacco use in dental caries development. Cent Eur J Public Health. 2007 Sep;15(3):116-21. doi: 10.21101/cejph.a3431. PMID 17958204
- [Result] Rooban T, Vidya K, Joshua E, Rao A, Ranganathan S, Rao UK, Ranganathan K. Tooth decay in alcohol and tobacco abusers. J Oral Maxillofac Pathol. 2011 Jan;15(1):14-21. doi: 10.4103/0973-029X.80032. PMID 21731272